CLINICAL TRIAL: NCT03962868
Title: Endoscopic Submucosal Dissection (ESD) Versus Endoscopic Mucosal Resection (EMR) for Large Non Pedunculated Colonic Adenomas: a Randomized Comparative Trial
Acronym: RESECT COLON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 87RI18_0002 (RESECT COLON)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colonic Polyp
Keywords: Colonic Polyp; large non pedunculated; colonic adenoma; Endoscopic submucosal dissection; Endoscopic Mucosal Resection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic submucosal dissection (ESD) (Experimental)
  Interventions: Procedure: Experimental procedure : ESD
- Endoscopic Mucosal Resection (WF-piece meal EMR) (Active Comparator)
  Interventions: Procedure: Comparison procedure: WF-piece meal EMR

INTERVENTIONS:
Procedure: Experimental procedure : ESD — ESD is a new endoscopic resection procedure that allows en-bloc resection for large superficial colorectal neoplasms. It used dedicated devices and consists in a deep submucosal dissection under the lesion after surelevation thanks to submucosal fluid injection and mucosal incision all around the lesion. The en bloc resection allows a perfect pathological analysis and a very low risk of recurrence (<1.5%)
  Arms: Endoscopic submucosal dissection (ESD)
Procedure: Comparison procedure: WF-piece meal EMR — WF-piece meal EMR is an older endoscopic resection technique. After surelevation of the lesion thanks to fluid submucosal injection, the precancerous lesion is resected in several pieces using a polypectomy snare. At the end of the procedure when macroscopically visible adenoma has been totally resected a snare tip coagulation of the margin of the scar is performed to destroy potential non visible residual adenoma. This procedure is quicker, safer than ESD but result in more recurrent disease (from 10 to 30% for lesions larger than 25 mm).
  Arms: Endoscopic Mucosal Resection (WF-piece meal EMR)

SUMMARY:
Initially developed in Japan for the treatment of endemic superficial gastric cancers, endoscopic submucosal dissection (ESD) allows resection of pre-neoplastic and neoplastic lesions of the digestive tract into a single fragment. It allows a perfect pathological analysis, and decreases the rate of recurrence of the adenoma to less than 2% However, this procedure, which is technically more challenging, is also more risky (perforation rate at 4% vs. 1% for WF-EMR) and longer. Submucosal dissection is also more expensive in terms of equipment, but this difference can be offset by the cost of the high number of iterative colonoscopies required in patients who have had endoscopic resection by WF-EMR.

Scientific debate is agitating the Western world1,2 and Japanese experts do not perform WF-EMR anymore, whereas no comparative prospective study has compared these two procedures.

We therefore propose to compare these two endoscopic resection strategies in terms of recurrence rate at 6 months and to estimate the differential cost-effectiveness and cost-utility ratios over a 36-month time horizon.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from non-pedunculated polyp suspected larger than 25 mm in the colon
* Colon localization beyond 15 cm of the anal margin.
* Indication for endoscopic treatment
* Patients aged ≥ 18 years old
* Patients able to fill in questionnaires written in French

Exclusion Criteria:

* Prior endoscopic resection attempt
* Contra-indication to colonoscopy
* Contra-indication to general anesthesia
* Inability to stop antiplatelet agents and anti-coagulant according to the European Society of Gastro-Intestinal Endoscopy guidelines.
* Recurrent adenoma: post-endoscopic or surgical resection
* Pregnant or lactating women
* Genetic polyposis (Familial Adenomatous Polyposis, Lynch Syndrome, Peutz-Jeghers Syndrome)
* Inability to provide informed consent
* Patient under legal protection and or deprived of liberty by judicial or administrative decision
* Patient already participating in an interventional clinical research protocol
* Patient who cannot be followed for the duration of the study
* Non-pedunculated polyp ≤ 25 mm
* More than one lesion > 25 mm that fulfilled the inclusion criteria
* Suspicion of deep submucosal cancer by analysis of macroscopic appearance (Paris 0-III), vascular pattern and pit pattern (SANO IIIB, KUDO Vn)
* Non granular pseudodepressed Laterally spreading tumors due to the high risk of nonvisible submucosal cancer
* Polyp involving the appendice deeply (type 2 or 3 of classification of Toyonaga)
* Polyp inside the ileo-caecal valvula
* Tattoing under the lesion
* Inflammatory Bowel Disease with expected fibrosis (Crohn disease or ulcerative colitis)
* Colon localization < 15 cm of the anal margin.
* Polyp invading a diverticulum
* Pedunculated polyp
* Absence of lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Compare recurrence rate at follow-up colonoscopy | Month 6
  Compare between two groups

SECONDARY OUTCOMES:
Proportion of R0 resection rate | Month 1
  Compare between two groups
Cumulative complications rate after treatment | Month 1
  Compare between two groups
Endoscopic curative resection rate without surgery | Month 36
  Compare between two groups
Quality of life over time | Month 36
  Compare between two groups at Month 1, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36
Cost-effectiveness ratio | Month 36
  Compare between two groups
Cost-utility ratio | Month 36
  Compare between two groups
Cumulative surgical referral rate | Month 36
  Compare between two groups
Compare the proportion of technical failure | Day 1
  Compare between two groups

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - University Hospital, Limoges, Limoges, France
  - Jean Mermoz Hospital, Lyon, France
  - Edouard Herriot Hospital, Lyon
  - Nancy University Hospital, Nancy
  - Cochin Hospital, Paris
  - Pontchaillou Hospital, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacques J, Schaefer M, Wallenhorst T, Rosch T, Lepilliez V, Chaussade S, Rivory J, Legros R, Chevaux JB, Leblanc S, Rostain F, Barret M, Albouys J, Belle A, Labrunie A, Preux PM, Lepetit H, Dahan M, Ponchon T, Crepin S, Marais L, Magne J, Pioche M. Endoscopic En Bloc Versus Piecemeal Resection of Large Nonpedunculated Colonic Adenomas : A Randomized Comparative Trial. Ann Intern Med. 2024 Jan;177(1):29-38. doi: 10.7326/M23-1812. Epub 2023 Dec 12. PMID 38079634